CLINICAL TRIAL: NCT00279435
Title: A Randomized, Double-blind, Multicenter Study of Visilizumab Versus Placebo in Subjects With Intravenous Steroid-refractory Ulcerative Colitis Previously Responsive in a Visilizumab Study
Brief Title: Study of Visilizumab Versus Placebo in Subjects With Intravenous Steroid-refractory Ulcerative Colitis Previously Responsive in a Visilizumab Study
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: company decision based on other studies
Sponsor: Facet Biotech (Industry)
Collaborators: PDL BioPharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 291-417
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-03

CONDITIONS: Ulcerative Colitis
Keywords: Intravenous, Steroid-Refractory, Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — visilizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: visilizumab
- visilizumab (Experimental)
  Interventions: Drug: visilizumab

INTERVENTIONS:
Drug: visilizumab

SUMMARY:
The purpose of this study is to compare the efficacy, safety, pharmacokinetics, and immunogenicity in subjects retreated with visilizumab or placebo after a response in a prior visilizumab study.

DETAILED DESCRIPTION:
The purpose of this study is to compare the efficacy, safety, pharmacokinetics, and immunogenicity in subjects retreated with visilizumab or placebo after a response in a prior visilizumab study.

PDL BioPharma, Inc. was formerly known as Protein Design Labs, Inc.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 years of age or older.
* Only 1 prior treatment course with visilizumab (or placebo in a blinded visilizumab study).
* Response (as defined in parent protocol) of intravenous steroid-refractory ulcerative colitis (IVSR-UC) disease to visilizumab or placebo.
* Symptomatic worsening (ie, an increase of ≥3 points in MTWSI score) from the subject's best response on the parent study, an MTWSI score of ≥9, sustained for at least 2 assessments performed at least 1 week apart, and a confirmatory MTWSI ≥8 within 1 day prior to randomization.
* CD4^+ T-cell count ≥ 200 cells/mcL at screening for this protocol, or ≥ 80% of the subject's screening baseline count prior to enrollment on the parent study.
* Mayo assessment (including flexible sigmoidoscopy) performed by a trained, blinded evaluating physician within 2 weeks prior to randomization.
* Adequate contraception from the day of consent through 3 months after the last dose of study drug.
* Negative serum pregnancy test.
* Negative Clostridium difficile test.
* Signed and dated informed consent, and Health Insurance Portability and Accountability Act (HIPAA) if applicable.

Exclusion Criteria:

* UC requiring immediate surgical, endoscopic, or radiologic interventions.
* White blood cell count less than 2.5 x 10^3/mcL; platelet count less than 150 x 10^3/mcL; or hemoglobin less than 8 g/dL.
* Active, medically significant infections, particularly those of viral etiology, eg, known cytomegalovirus (CMV) colitis. This includes any incidence of opportunistic infections within the past 12 months.
* Live vaccination within 6 weeks prior to randomization.
* Significant organ dysfunction, including cardiac, renal, liver, CNS, pulmonary, vascular, gastrointestinal, endocrine, or laboratory abnormality, history of myocardial infarction, coronary artery disease, congestive heart failure, or arrhythmias within 6 months prior to consent.
* History of lymphoproliferative disorder (LPD) or malignancy other than nonmelanoma skin cancer or carcinoma in situ of the cervix that has been adequately treated within the past five years.
* Seropositive for infection with human immunodeficiency virus (HIV-1), hepatitis B virus (HBV) surface antigen, or hepatitis C virus (HCV).
* Pregnancy or nursing.
* Treatment with any other UC salvage drugs (including but not limited to infliximab or another anti-TNF-a drug, cyclosporine, tacrolimus [FK506], adalimumab, thalidomide, or another experimental agent), or therapies (surgery, pheresis, affinity columns) since the first course of treatment with study drug in the parent visilizumab study.
* Treatment with any other investigational drug or therapy within 60 days prior to randomization.
* Nontherapeutic levels of chronic antiseizure medications in subjects with a history of seizures.
* Any condition that, in the investigator's opinion, makes the subject unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-08; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (39):
- United States (9):
  - Atlanta, Georgia
  - Louisville, Kentucky
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - New York, New York
  - Hershey, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Nashville, Tennessee
  - Murray, Utah
- Australia (4):
  - Box Hill, Victoria
  - Fremantle
  - Herston
  - Liverpool
- Vienna, Austria
- Belgium (2):
  - Ghent
  - Leuven
- Canada (3):
  - Winnipeg, Manitoba
  - Hamilton, Ontario
  - Calgary
- Croatia (2):
  - Osijek
  - Zagreb
- Czechia (2):
  - Brno
  - Prague
- France (3):
  - Clichy
  - Lille
  - Paris
- Germany (3):
  - Berlin
  - Freiburg im Breisgau
  - Kiel
- Hungary (4):
  - Csabai Kapu
  - Szekszárd
  - Vasvári Pál
  - Vác
- Tel Litwinsky, Israel
- Bologna, Italy
- Amsterdam, Netherlands
- Norway (2):
  - Oslo
  - Tromsø
- Odesa, Ukraine